CLINICAL TRIAL: NCT06782594
Title: A Multicenter, Randomized, Double-blind, Parallel, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy of Mosapride Citrate Injection in the Treatment of Postoperative Gastrointestinal Dysfunction
Brief Title: A Phase Ⅱ Study of Mosapride Citrate Injection in the Treatment of Postoperative Gastrointestinal Dysfunction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTP-MSBL-003
Record Dates: First submitted 2025-01-08; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Gastrointestinal Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mosapride Citrate Injection(low) (Experimental): Mosapride Citrate Injection, iv, 4mg, bid, for 3 to 5 days
  Interventions: Drug: Mosapride Citrate Injection(low)
- Mosapride Citrate Injection(high) (Experimental): Mosapride Citrate Injection, iv, 8mg, bid, for 3 to 5 days
  Interventions: Drug: Mosapride Citrate Injection(high)
- Placebo (Placebo Comparator): Placebo, iv, bid, for 3 to 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mosapride Citrate Injection(high) — Mosapride Citrate Injection, iv, 8mg, bid, for 3 to 5 days
  Arms: Mosapride Citrate Injection(high)
Drug: Mosapride Citrate Injection(low) — Mosapride Citrate Injection, iv, 4mg, bid, for 3 to 5 days
  Arms: Mosapride Citrate Injection(low)
Drug: Placebo — Placebo, iv, bid, for 3 to 5 days
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, parallel, placebo-controlled phase II clinical study.

DETAILED DESCRIPTION:
The study was divided into three phases: screening period (within 28 days before surgery), treatment period (3-5 days), and follow-up period (7 days after the last dose). Subjects entered the screening period after signing the informed consent form. Subjects who met the inclusion criteria and those who did not meet the exclusion criteria were randomly assigned to trial group 1, trial group 2, or control group at a random ratio of 1:1:1, and received mosapride citrate injection or placebo, respectively. After the treatment period, the subjects entered the follow-up period after the treatment ended.

ELIGIBILITY:
Inclusion Criteria:

1）Voluntary participation and signing of informed consent;

2) Aged ≥18 years and ≤75 years and BMI≤28kg/m2, regardless of gender;

3) Patients undergoing elective laparoscopic-assisted intestinal resection and the surgical site is part of the intestinal segment from the ileocecal region to the sigmoid colon;

4) Vital organ functions meet the following requirements:iver function:

ALT and AST≤3×ULN, total bilirubin level≤2×ULN;

Renal function: serum creatinine (Cr)≤1.5×ULN or creatinine clearance≥50mL/min (when Cr>1.5×ULN);

Blood routine examination: hemoglobin (HGB)≥80g/L;

Blood biochemistry: albumin (ALB)≥30g/L;

5) Those classified as physical condition 1 to 3 by the American Society of Anesthesiologists (ASA).

Exclusion Criteria:

1) Patients with a history of clinically significant drug allergy or known allergy to the study drug ingredients and excipients;

2）Those who have a history of severe heart, lung, liver, kidney, blood, endocrine, immune, skin, neurological or mental diseases in the past two years or currently have diseases of the above systems;

3) Those with a history of drug abuse in the past 6 months;

4) Those with a history of constipation in the past 6 months (less than 3 bowel movements per week);

5) Severe mechanical intestinal obstruction that is not expected to be relieved after surgery, short bowel syndrome, significant gastrointestinal motility disorders (such as gastroparesis, scleroderma, chronic intestinal pseudo-obstruction), poorly controlled Those with diabetes (HbA1c>8.5%) or gastrointestinal pacemakers installed in their bodies;

6) Patients with inflammatory bowel disease (ulcerative colitis or Crohn's disease) and intestinal adhesions;

7) Those who have undergone major abdominal surgery (such as gastrectomy, gastric bypass, sleeve gastrectomy, gastric band surgery, Whipple surgery, pancreatectomy, colectomy, hemicolectomy);

8) QTcF interval: ≥450 milliseconds for men and ≥470 milliseconds for women (the QT interval must be corrected for heart rate using the Fridericia formula [QTcF]);

9) Patients who received chemotherapy within 4 weeks before surgery;

10) Those who are scheduled for emergency surgery or undergo any of the following surgeries: appendectomy, low anterior resection, colostomy, ileostomy, or stoma reversal, or diagnosed with needing proctocolectomy/low anterior resection Subjects whose disease may cause impaired rectal function or postoperative incontinence (except for lesions that do not involve the sigmoid colon and above);

11) Within 3 days before the first dose, patients had received stimulants such as alvimopan, erythromycin, prucalopride, metoclopramide, domperidone, cisapride, mosapride, renzapride or azithromycin. Gastrointestinal motility drugs;

12) Pregnant or lactating women, as well as those who plan to become pregnant or donate sperm or eggs during the study period and within 3 months after the end of the study, and are unwilling to use a medically recognized contraceptive measure (such as intrauterine contraceptive device or contraceptive) during the study period. sets);

13) Participated in other clinical trials within 3 months before enrollment;

14) Other subjects deemed unsuitable for inclusion by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The time to first flatus recorded by postoperative patients | up to 3 to 5 days
  Comparison of the effects of experimental drugs and placebo on the time to first flatus postoperative patients

CONTACTS AND LOCATIONS:
Overall Officials: Guihua Wang, MD, Principal Investigator — TONGJI HOSPITAL AFFILIATED TO TONGJI MEDICAL COLLEGE HUST
Locations (2):
- China (2):
  - Shandong New Time Pharmaceutical Co., LTD, Feixian, Shandong
  - Tongji Hospital Affiliated to Tongji Medical College Hust, Wuhan